CLINICAL TRIAL: NCT04244682
Title: Brain Stimulation Study of Human Cognition Using Repetitive Transcranial Magnetic Stimulation (rTMS)
Brief Title: rTMS Brain Stimulation and Cognition
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment and enrollment were suspended due to COVID-19 and ultimately the study was withdrawn due trained personnel moving on to new projects.
Sponsor: Stephan Hamann (Other)
Responsible Party: Sponsor-Investigator, Stephan Hamann, Professor, Emory University
Organization: Emory University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00115488
Record Dates: First submitted 2020-01-27; First posted 2020-01-28 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Episodic Memory Retrieval
Keywords: Imaging; Neuroanatomy; Magnetic Resonance Imaging (MRI); Neuroscience
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Healthy participants receiving rTMS (Other): Participation will require up to three visits. One visit will take up to an hour, and the other visits will each take up to three hours each. During the first visit, participants will be consented, and their brains will be scanned using magnetic resonance imaging. Participants will receive rTMS during two study visits.
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — In the rTMS procedure a small plastic coil will be placed next to the participant's head. The position of the coil will be guided by neuro-navigational software utilizing the individual's MRI scan. The coil will be placed over the relevant brain region using the Brainsight TMS-MRI co-registration system for visualizing the coil position with respect to the participant's individual MRI scan. The coil will then generate a series of repetitive magnetic pulses, and stimulation will occur, disrupting typical function of the targeted brain region.

SUMMARY:
This study will use repetitive transcranial magnetic stimulation (rTMS) (a way to use a powerful magnet to cause temporary impairment to the function of a brain region) to test whether certain parts of the brain are necessary to various aspects of memory and emotion. Participation will require up to three visits. One visit will take up to an hour, and the other visits will each take up to three hours each. During the first visit, participants will be consented, and their brains will be scanned using magnetic resonance imaging.

DETAILED DESCRIPTION:
Memory and emotion are complex cognitive processes. To understand memory and emotion better, it is helpful to break them down into component processes and examine how each of these component processes is supported by brain. One way to do this is to safely and reversibly impair the function of a brain region that are believed to support some of these component processes and observe changes in behavior.

A high-resolution three-dimensional image of a participant's brain will be created using magnetic resonance imaging (MRI) scanning (about 10 minutes in the scanner). Either the same day or on a following day, participants will return and will be exposed to emotional and/or neutral stimuli. Either before or after being exposed to the stimuli, the participants will have their brain mildly stimulated using rTMS. This stimulation will be at or below the levels which the FDA has deemed safe for treatment of depression, and will temporarily reduce brain activity in the targeted area. The behavior of the participant's memory, emotional processing, or related cognitive functions will be tested by asking them questions about emotional and/or neutral stimuli. Depending on which condition the participant is part of, the researchers may then bring the participant back, and repeat this procedure on a different day stimulating another brain region.

Up to 80 participants will be identified via word of mouth, the psychology department research pool, and via flyers posted on Emory campus. Participants will give informed consent to participate and will be compensated for their time.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* healthy

Exclusion Criteria:

* personal or first-degree family history of epileptic seizure
* a known brain injury
* claustrophobia
* taking certain medications that may increase the risk of seizures (e.g., bupropion, varenicline, chlorpromazine, theophylline) or reduce the effects of rTMS, such as benzodiazepines
* current use of medication for neurological or psychiatric conditions
* internal metallic implant, device, or foreign body
* left handedness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change in Remember/Familiar Scale Score | Day 1 (first rTMS visit), Up to Day 14 (second rTMS visit)
  Memory accuracy will be assessed using a remember/familiar scale that was created for this study, based on common scales used in basic memory research. This instrument is a a 3-option categorical forced-choice self-report measure that assesses the accuracy of a participant's memory for an item. This measure assesses whether the participant has no conscious memory of the item (New), whether they have a specific conscious recollection of having seen the item before (Remember), or whether they have a conscious sense of having seen the item before but they cannot recollect any specific details relating to the item (Familiar). This scale will be scored by calculating the number of Hits (old items endorsed as remembered/familiar), Misses (old items endorsed as new), Correct Rejections (new items endorsed as new), and False Alarms (new items endorsed as familiar/remembered), and then calculating a sensitivity index (d') for each participant.
Change in Confidence Scale Score | Day 1 (first rTMS visit), Up to Day 14 (second rTMS visit)
  Memory confidence will be assessed using a confidence scale that was created for this study, based on common scales used in basic memory research. The confidence scale is a 4-point ordinal forced-choice self-report measure that assess the subjective confidence a participant feels in their memory for an item. The scale's choices are 1 = Little Confidence, 2 = Some Confidence, 3 = Moderate Confidence, and 4 = High Confidence. The scale's responses will be averaged for each participant.
Change in Vividness Scale Score | Day 1 (first rTMS visit), Up to Day 14 (second rTMS visit)
  Memory vividness will be assessed using a vividness scale that was created for this study, based on common scales used in basic memory research. The vividness scale is a 4-point ordinal forced-choice self-report measure that assess the subjective vividness a participant experiences of their memory for an item. The scale's choices are 1 = Not Vivid, 2 = Slightly Vivid, 3 = Moderately Vivid, and 4 = Highly Vivid. The scale's responses will be averaged for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Hamann, PhD, Principal Investigator — Emory University

IPD SHARING:
Plan to Share IPD: No